CLINICAL TRIAL: NCT04503746
Title: A Multi-center, Randomized, Double-Blind, Phase II Clinical Trial to Evaluate the Efficacy and Safety of 12-week Treatment of ALH-L1005 600 mg or 1200 mg in Patients With Chronic Periodontitis
Brief Title: A Study to Evaluate the Efficacy and Safety of ALH-L1005 in Patients With Chronic Periodontitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AngioLab, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AL102-PDT
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Chronic Periodontitis
Keywords: periodontitis
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo twice a day
  Interventions: Drug: Placebo
- ALH-L1005 600 mg (Experimental): ALH-L1005 300 mg twice a day
  Interventions: Drug: ALH-L1005 600mg/day
- ALH-L1005 1,200 mg (Experimental): ALH-L1005 600 mg twice a day
  Interventions: Drug: ALH-L1005 1,200mg/day

INTERVENTIONS:
Drug: ALH-L1005 600mg/day — ALH-L1005 300mg 2 tablet and placebo 2 tablet
  Arms: ALH-L1005 600 mg
Drug: ALH-L1005 1,200mg/day — ALH-L1005 300mg 4 tablet
  Arms: ALH-L1005 1,200 mg
Drug: Placebo — Placebo 4 tablet
  Arms: Placebo

SUMMARY:
The main objective of this study is to evaluate efficacy and safety of ALH-L1005 in patients with chronic periodontitis

ELIGIBILITY:
Inclusion Criteria:

* Men or women ages 18 and over, under 79 years of age
* Patients diagnosed with chronic periodontitis
* Patients with 4 teeth and over whose pocket depth is ≥ 4 mm and clinical attachment level is ≥ 3 mm
* Patients who are voluntarily participated in clinical trial

Exclusion Criteria:

* History of antibiotic therapy within the 1 month prior to study
* Those who had undergone any dental surgical or non-surgical therapy within 3 months prior to the start of the study
* Subjects who are pregnant/ lactating
* Smokers
* Patients who take Anticoagulants or Antiplatelet Agents
* With Systemic diseases that affect periodontal conditions such as: diabetes, hypertension and diseases of immune system

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Change in Pocket Depth(PD) | baseline, 12 weeks
  Change in Pocket Depth in Subjects

SECONDARY OUTCOMES:
Change in Pocket Depth(PD) | baseline, 4 weeks, 8 weeks
  Change in Pocket Depth in Subjects
Change in Clinical Attachment Level(CAL) | baseline, 4 weeks, 8 weeks, 12 weeks
  Change in Clinical Attachment Level in Subjects
Change in Gingival recession(GR) | baseline, 12 weeks
  Change in Gingival recession in Subjects
Change in Bleeding on probing(BOP) score | baseline, 12 weeks
  Change in Bleeding on probing score in Subjects

CONTACTS AND LOCATIONS:
Locations (1):
- AngioLab, Inc., Daejeon, Daejeon Gwangyeogsi, South Korea

IPD SHARING:
Plan to Share IPD: No